CLINICAL TRIAL: NCT00754988
Title: A Multicenter, Randomized, Double-dummy, Placebo and Active-controlled Study to Assess the Safety, Tolerability and Effect of Taspoglutide on Glycemic Control Compared to Sitagliptin and Placebo in Patients With Type II Diabetes Mellitus Inadequately Controlled With Metformin.
Brief Title: A Study of Taspoglutide Versus Sitagliptin for the Treatment of Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC21713; 2008-001854-42
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Sitagliptin Phosphate; taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Once daily oral administration of placebo (matching sitagliptin). Once weekly sc injection of placebo (matching taspoglutide). Continued treatment with metformin at prescribed doses.
  Interventions: Drug: Metformin; Drug: Placebo (matching sitagliptin); Drug: Placebo (matching taspoglutide)
- Sitagliptin (Active Comparator): Once daily oral administration of 100 mg of sitagliptin. Once weekly sc injection of placebo (matching taspoglutide). Continued treatment with metformin at prescribed doses.
  Interventions: Drug: Metformin; Drug: Placebo (matching taspoglutide); Drug: Sitagliptin
- Taspoglutide 10 mg (Experimental): Once weekly subcutaneous (sc) injection of 10 mg of taspoglutide. Once daily oral administration of placebo (matching sitagliptin). Continued treatment with metformin at prescribed doses.
  Interventions: Drug: Metformin; Drug: Placebo (matching sitagliptin); Drug: Taspoglutide
- Taspoglutide up-titrated to 20 mg (Experimental): Once weekly sc injection of 10 mg of taspoglutide for the first 4 weeks, then up-titrated to once weekly sc injection of 20 mg of taspoglutide from week 5 onwards. Once daily oral administration of placebo (matching sitagliptin). Continued treatment with metformin at prescribed doses.
  Interventions: Drug: Metformin; Drug: Placebo (matching sitagliptin); Drug: Taspoglutide

INTERVENTIONS:
Drug: Metformin — As prescribed
Drug: Placebo (matching sitagliptin) — Once daily oral administration of placebo (matching sitagliptin).
  Arms: Placebo; Taspoglutide 10 mg; Taspoglutide up-titrated to 20 mg
Drug: Placebo (matching taspoglutide) — Once weekly subcutaneous (sc) injection of placebo (matching taspoglutide).
  Arms: Placebo; Sitagliptin
Drug: Sitagliptin — Once daily oral administration of 100 mg of sitagliptin.
  Arms: Sitagliptin
Drug: Taspoglutide — Once weekly subcutaneous (sc) injection of 10 mg or 20 mg of taspoglutide.
  Arms: Taspoglutide 10 mg; Taspoglutide up-titrated to 20 mg

SUMMARY:
This 4 arm study will assess the efficacy, safety and tolerability of taspoglutide compared to sitagliptin and placebo in patients with type 2 diabetes mellitus inadequately controlled with metformin. Patients will be randomized to receive taspoglutide (10mg once weekly or 10mg once weekly for 4 weeks followed by 20mg once weekly), sitagliptin 100mg once daily or placebo, in a ratio of 2:2:2:1, in addition to their continued prestudy metformin treatment. After 24 weeks of treatment, patients on active treatment will continue on the same treatment and patients on placebo will be switched to taspoglutide 10mg once weekly or taspoglutide 20mg once weekly (after 4 weeks of taspoglutide 10mg once weekly). The anticipated time on study treatment is 2+ years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes receiving metformin (>=1500mg/day) for at least 12 weeks;
* HbA1c >=7.0% and <=10.0% at screening;
* BMI >=25 (>23 for Asians) and <=45kg/m2 at screening;
* stable weight +/- 5% for at least 12 weeks prior to screening.

Exclusion Criteria:

* history of type 1 diabetes mellitus or acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma in the previous 6 months;
* evidence of clinically significant diabetic complications;
* clinically symptomatic gastrointestinal disease;
* myocardial infarction, coronary artery bypass surgery, post-transplantation cardiomyopathy or stroke within the previous 6 months;
* known hemoglobinopathy or chronic anemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Mean changes in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose; change from baseline in body weight; responder rates for HbA1c (target <=7.0%, <=6.5%); responder rates for body weight; change from baseline in lipid profile; beta cell function. | 24 weeks
Safety: Adverse events, vital signs, physical examination, clinical laboratory tests, ECG and anti-taspoglutide antibodies. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (136):
- United States (61):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Tallassee, Alabama
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Huntington Beach, California
  - La Jolla, California
  - Los Angeles, California
  - Roseville, California
  - San Francisco, California
  - Tacoma, California
  - Colorado Springs, Colorado
  - New London, Connecticut
  - Manati, District of Columbia
  - Daytona Beach, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Panama City, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Conyers, Georgia
  - Snellville, Georgia
  - Honolulu, Hawaii
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - South Bend, Indiana
  - Baltimore, Maryland
  - Brockton, Massachusetts
  - Cadillac, Michigan
  - Brooklyn Center, Minnesota
  - Minneapolis, Minnesota
  - City of Saint Peters, Missouri
  - Fulton, New York
  - Hudson, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Shelby, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Delaware, Ohio
  - Marion, Ohio
  - Corvallis, Oregon
  - Eugene, Oregon
  - Aliquippa, Pennsylvania
  - Beaver, Pennsylvania
  - Erie, Pennsylvania
  - Reading, Pennsylvania
  - Shippensburg, Pennsylvania
  - Warminster, Pennsylvania
  - Anderson, South Carolina
  - Kingsport, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - South Burlington, Vermont
  - Hampton, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Federal Way, Washington
- Argentina (2):
  - Buenos Aires
  - Mar del Plata
- Australia (2):
  - Freemantle, Queensland
  - Adelaide, South Australia
- Canada (5):
  - London, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
- France (5):
  - Bondy
  - Nantes
  - Poitiers
  - Rennes
  - Saint-Mandé
- Germany (7):
  - Berlin
  - Dormagen
  - Dresden
  - Kiel Kronshagen
  - München
  - Sulzbach-Rosenberg
  - Villingen-Schwenningen
- Larissa, Greece
- Mexico (6):
  - Cuernavaca
  - Hermosillo
  - Jalisco
  - Mexico City
  - Monterrey
  - Pachuca
- Norway (2):
  - Elverum
  - Oslo
- Lima, Peru
- Poland (7):
  - Bialystok
  - Gdansk
  - Kamieniec Ząbkowicki
  - Rzeszów
  - Skierniewice
  - Sobótka
  - Wroclaw
- Puerto Rico (2):
  - Caguas
  - Carolina
- Romania (4):
  - Bucharest
  - Buzău
  - Cluj-Napoca
  - Ploieşti
- Slovakia (5):
  - Levice
  - Prešov
  - Šamorín
  - Trebišov
  - Trenčín
- South Africa (2):
  - Cape Town
  - Pretoria
- South Korea (3):
  - Gyeonggi-do
  - Seoul
  - Wŏnju
- Spain (4):
  - Bacarot Alicant, Alicante
  - Almería, Almeria
  - Seville, Sevilla
  - Valencia, Valencia
- Sweden (3):
  - Ljungby
  - Örebro
  - Stockholm
- Switzerland (3):
  - Basel
  - Geneva
  - Zurich
- Taiwan (3):
  - Taichung
  - Taipei
  - Taoyuan
- Thailand (2):
  - Bangkok
  - Songkhla
- Istanbul, Turkey (Türkiye)
- United Kingdom (5):
  - Bexhill-on-Sea
  - Crawley
  - Glasgow
  - Hinckley
  - Reading